CLINICAL TRIAL: NCT01654913
Title: Influence of the Inspired Oxygen Fraction on the Noninvasive Measurement of Hemoglobin Using Two Different Devices (Namely Pronto 7 and NBM-200)
Brief Title: Influence of Oxygen on Non-invasive Measurement of Hemoglobin
Acronym: Hb-O2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/16; 2012-A00416-37 (Other: ANSM)
Record Dates: First submitted 2012-07-16; First posted 2012-08-01 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Anesthesia
Keywords: hemoglobin determination; oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- surgical patients (Experimental): patients studied just before induction of anesthesia
  Interventions: Device: hemoglobin measurement

INTERVENTIONS:
Device: hemoglobin measurement — Non invasive hemoglobin measurements (Pronto 7 device and NBM-200 device)will be made with :
  * at baseline (simultaneous blood sample for a laboratory measurement of hemoglobin),
  * with the patient breathing oxygen via a face-mask (FiO2 50 ± 5%),
  * with the patient breathing oxygen via a face-mask (FiO2 90 ± 5%) (simultaneous blood sample for a laboratory measurement of hemoglobin).

SUMMARY:
This study examines the effect of oxygen supplementation on the non-invasive measurement of hemoglobin.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for a potentially hemorrhagic surgical procedure

Exclusion Criteria:

* anomaly (malformation, infection, swelling, irritation, ulceration, degenerative changes or significant edema) of the fingers,
* tremors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
influence of the inspired oxygen fraction on the noninvasive measurement of hemoglobin (Pronto 7 and NBM-200 devices) | one year (end of the recrutement period)
  Statistical comparison of the 3 measurements (baseline, FiO2 50%, FiO295%) for each device

SECONDARY OUTCOMES:
agreement between the noninvasive methods of measurement of hemoglobin and the laboratory analysis | one year (end of the recrutement period)
  Statistical comparison of the 2 devices

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital Lariboisière, Paris
  - Hopital Foch, Suresnes

REFERENCES:
- [Background] Gayat E, Aulagnier J, Matthieu E, Boisson M, Fischler M. Non-invasive measurement of hemoglobin: assessment of two different point-of-care technologies. PLoS One. 2012;7(1):e30065. doi: 10.1371/journal.pone.0030065. Epub 2012 Jan 6. PMID 22238693
- [Background] Gayat E, Bodin A, Fischler M. Instability in non-invasive haemoglobin measurement: a possible influence of oxygen administration. Acta Anaesthesiol Scand. 2011 Aug;55(7):902. doi: 10.1111/j.1399-6576.2011.02469.x. Epub 2011 Jun 9. No abstract available. PMID 21658016
- [Derived] Gayat E, Imbert N, Roujansky A, Lemasle L, Fischler M. Influence of Fraction of Inspired Oxygen on Noninvasive Hemoglobin Measurement: Parallel Assessment of 2 Monitors. Anesth Analg. 2017 Jun;124(6):1820-1823. doi: 10.1213/ANE.0000000000001783. PMID 28221201